CLINICAL TRIAL: NCT07033338
Title: The Effect of Occupational Activities and Finger Exercise Program on Hand Grip Strength and Activities of Daily Living in Elderly Individuals With Dementia: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emel Dogan (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Emel Dogan, Doctoral Student, Department of Nursing, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Selcuk.Emel.01
Record Dates: First submitted 2025-04-07; First posted 2025-06-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Aged 65 Years or Older; Cognitive Decline; Dementia
Keywords: Finger exercise; Elderly; Occupational activities; Hand grip strength; Activities of daily living; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group was composed of elderly individuals aged 65 years and older who were residing in a nursing home and were not bedridden The intervention group was composed of elderly individuals aged 65 years and older who were residing in a nursing home and were not bedridden. A total of 25 out of 50 participants were randomly assigned to this group. The intervention included a structured program of occupational activities and finger exercises implemented 3 days per week for 8 weeks, aiming to improve hand grip strength and activities of daily living. The intervention was delivered by trained healthcare staff, and informed consent was obtained from all participants.
  Interventions: Behavioral: Occupational Activities and Finger Exercise Program
- Control Group (No Intervention): The control group consisted of elderly individuals aged 65 years and older who were residing in a nursing home and were not bedridden. A total of 25 out of 50 participants were randomly assigned to this group. Participants in this group did not receive any intervention and continued with their usual care routines. They were evaluated at the same time points as the intervention group to compare outcomes such as hand grip strength and daily living activities.

INTERVENTIONS:
Behavioral: Occupational Activities and Finger Exercise Program — The intervention group received the program three days a week (Wednesday, Thursday, and Friday), once daily, with sessions held from 10:00 to 12:00 in the morning and from 14:00 to 16:00 in the afternoon. The participants were divided into two subgroups (13 participants in the first group, 12 in the second). The intervention consisted of a combined occupational activities and finger exercise program. Each session began with finger exercises, followed by occupational activities. The finger exercises involved movements requiring the participation of the fingers, hands, and arms, and were performed in 10 progressive steps. These movements were designed to promote engagement without causing fatigue or discomfort in elderly participants. Occupational activities included threading beads, completing line patterns, sewing buttons, assembling wooden blocks, performing cutting exercises, limited painting, dough manipulation, cutting and gluing, wrapping rope, tying rope between two points, stack
  Arms: Intervention Group

SUMMARY:
As people age, cognitive functions, muscle mass, and hand strength tend to decrease. Reduced hand grip strength in the elderly can make it harder for them to perform daily tasks such as buttoning clothes, pulling zippers, or opening doors. These difficulties can lead to a reduced quality of life and increased need for assistance and institutional care. Activities of daily living (ADL) are a key indicator of an older adult's ability to live independently.

This study aimed to examine whether an occupational activities and finger exercise program helps improve hand grip strength and the ability to perform daily tasks among older adults with mild dementia. The program includes hand and finger exercises combined with creative and functional tasks such as sewing, painting, and using tools. Supporting physical and cognitive function through such activities may help improve the independence and well-being of elderly individuals living in institutions.

DETAILED DESCRIPTION:
The study was planned as a randomized, parallel-group experimental design. It was conducted in Konya Dr. İsmail Işık Nursing Home. Fifty randomly selected individuals who were over 65 years of age, not bedridden, and who agreed to participate voluntarily were included in the study.

Pre-tests After the individuals included in the study group were informed about the study and gave their consent, pre-test applications (information form, Barthel Index, and hand and finger grip strength measurement) were performed. The hand and finger grip strength measurements and data collection were performed by an independent physiotherapist who was experienced in this field. The measurements and data collection were performed in the rooms of elderly individuals with dementia who stayed in a private room, while others were evaluated in a separate room.

Post-tests Post-tests (Barthel Index and hand and finger grip strength measurements) were carried out at the end of the 8th week by the same independent physiotherapist. The post-tests were also performed in the rooms of elderly individuals who stayed in a private room, while the others were in a separate room.

Intervention A pastime activities and finger exercise program was applied to the experimental group 3 times a week for 8 weeks. At the end of the program, post-test evaluations for hand grip strength and daily life activities in both the experimental and control groups were performed simultaneously. The data obtained as a result of the measurements - numbers, percentages, mean, minimum and maximum values - were analyzed using the independent groups t-test, Mann-Whitney U test, Wilcoxon test, and Shapiro-Wilk test for normal distributions. Ethics committee approval and institutional permission have been obtained for the study.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of dementia (MMSE score between 18-23)
* Age 65 years or older
* Not bedridden Exclusion Criteria
* Advanced osteoarthritis or neurological disorders
* Significant visual/hearing impairment interfering with communication
* Severe depression or behavioral disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Measurement of hand and finger grip strength in elderly individuals using digital dynamometer | Baseline and at 2 months (post-test)
  Hand grip strength was assessed using a digital hand dynamometer to evaluate upper extremity muscle performance. The test was performed on the dominant hand while the participant was in a seated position with the elbow flexed at 90 degrees. Three attempts were recorded, and the highest value (in kg) was used in the analysis.A pinchmeter is used to measure finger grip strength. Finger grip strength measurement should be performed while the individual is sitting on a chair, in the standard position recommended by the American Society of Hand Therapists (AETD); sitting position, shoulder adduction and elbow 90° flexion. In the test procedure, 3 measurements should be taken for finger grip strength with one minute intervals between each measurement and the averages should be recorded (American Society of Hand Therapists). Measurements were taken at baseline (prior to the intervention) and after 8 weeks of intervention.
Activities of Daily Living (ADL) - Standardized Questionnaire | Baseline and at 2 months (post-test)
  The level of independence in performing activities of daily living (ADL) was assessed using the Barthel Index. The aim was to assess the functional performance of elderly individuals in both the intervention and control groups. The difference in ADL scores between the groups was analyzed to determine the effect of the occupational activity and finger exercise program on daily living functions. Assessments were conducted at baseline and 8 weeks after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yeter Kitis, Professor, Principal Investigator — Gazi University Faculty of Nursing
Locations (1):
- Konya Dr. İsmail Işık Nursing Home, Konya, Meram/Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.